CLINICAL TRIAL: NCT06268197
Title: Feasibility and Acceptability of Interoception-Based Yoga for Chronic Pain
Brief Title: Interoception-Based Yoga for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0329
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Yoga Intervention (Experimental): Interoception-based yoga intervention, 2x/week for 6 weeks.
  Interventions: Behavioral: Yoga Intervention

INTERVENTIONS:
Behavioral: Yoga Intervention — The yoga intervention will consist of twice weekly, in-person, gentle Hatha yoga classes delivered by a certified yoga instructor. Each class will last 60-75 minutes and will include an introduction to the day's topic, an opening breathing/meditation practice, yoga postures, a closing breathing/meditation practice, and end with a savasana pose and intention setting for a home practice.

SUMMARY:
The purpose of this research is to examine the feasibility and acceptability of an interoception-based yoga program for chronic pain. Interoception involves your ability to feel sensations in your body (such as your heartbeat or muscle tension) as well as how you think about and interpret those sensations. Interoception may be an important component of chronic pain and the research team is studying whether yoga can change how you feel, think about, and interpret sensations in your body.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported chronic pain lasting ≥ 3 months (such as widespread musculoskeletal pain, fibromyalgia, migraine etc.)
* In the past week, has pain interfered with your day-to-day activities? Yes
* Self-reported ambulatory ability without an assistive device
* Self-reported ability to get on and off the floor without assistance.
* No ongoing mind-body practice (<1x/week over the past 6 months).
* Physical Activity Readiness Questionnaire Screen Pass or Physician Consent
* English-speaking
* Able and willing to provide consent
* No plans to move or travel outside the area in the next 2 months

Exclusion Criteria:

* Ages <18 or ≥ 65 at time of screening
* Pain lasting < 3 months
* In the past week, has pain interfered with your day-to-day activities? No
* Use of any assistive device (e.g. cane, walker, wheelchair).
* Inability to get on and off the floor without assistance.
* A consistent ongoing mind-body practice (mindfulness, yoga, meditation, tai chi, qigong), at least 1x/week over the past 6 months
* Physical Activity Readiness Questionnaire Screen Fail or non-consent of physician
* Non-English speaking
* Non-consent
* Plans to move or significant travel outside the area in the next 2 months
* Known pregnancy
* Recent surgery or acute bone, joint or nerve injury (within the past 6 months)
* Severe or progressive neurological conditions such as Parkinson's disease, dementia, multiple sclerosis, or acquired brain injury
* Separate pain-related diagnoses: cancer-related pain, complex regional pain syndrome, postural orthostatic tachycardia syndrome, functional neurological/ movement disorders
* Active or planned worker's compensation or personal injury claim
* Concurrent participation in another interventional study (e.g. physical activity, mind-body or drug trials)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Feasibility | Primary endpoint: 6 weeks
  Defined as achieving the target recruitment sample (N=25) in a 9-month period, 80% retention (N=20), 70% attendance rate, 70% home practice adherence and no serious adverse events.
Acceptability | Primary endpoint: 6 weeks
  Defined as >5/7 on acceptability questionnaire (1 = unacceptable, 7 = very acceptable)

SECONDARY OUTCOMES:
Interoceptive Sensibility | Primary endpoint: 6 weeks
  Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). Will take the mean of 5 MAIA-2 Subscales: attention regulation, emotional awareness, self-regulation, body listening, and trusting as the primary measure of preliminary efficacy. Planned post-hoc analyses will evaluate differential changes in all 8 subscales.
PROMIS Pain Interference | Primary endpoint: 6 weeks
  Short Form 8a

OTHER OUTCOMES:
Interoceptive Accuracy | Primary endpoint: 6 weeks
  Heartbeat Tracking Task
Mindfulness | Primary endpoint: 6 weeks
  Five Facet Mindfulness Questionnaire (FFMQ), planned covariate for interoceptive sensibility
PROMIS Pain Intensity | Primary endpoint: 6 weeks
  Short Form 3a, planned covariate for pain interference.
Quality of Life | Primary endpoint: 6 weeks
  36-Item Short Form Health Survey (SF-36)
Spiritual Wellbeing | Primary endpoint: 6 weeks
  Functional Assessment of Chronic Illness Therapy - Spiritual Wellbeing Scale (FACIT-Sp12)
Pain Impact | Primary endpoint: 6 weeks
  ASCQ Pain Impact Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Neha P Gothe, PhD, Principal Investigator — University of Illinois Urbana-Champaign; Steven Petruzzello, PhD, Principal Investigator — University of Illinois Urbana-Champaing
Locations (1):
- University of Illinois Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Voss S, Patel I, Skowron C, Petruzzello S, Gothe NP. Interoception-Based Yoga for Chronic Pain: A Pilot Feasibility Study. Glob Adv Integr Med Health. 2025 Nov 20;14:27536130251400362. doi: 10.1177/27536130251400362. eCollection 2025 Jan-Dec. PMID 41282370